CLINICAL TRIAL: NCT00001933
Title: Nefiracetam Therapy of Alzheimer's Type Dementia
Brief Title: Nefiracetam in the Treatment of Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 990139; 99-N-0139; NCT00000186 (obsolete NCT alias)
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2002-01

CONDITIONS: Alzheimer's Disease
Keywords: Acetylcholine; Clinical Trial; GABA; Cognition; Nicotine
MeSH Terms: conditions — Alzheimer Disease | interventions — nefiracetam

INTERVENTIONS:
Drug: Nefiracetam

SUMMARY:
Some of the thinking difficulties of Alzheimer's patients may be due to a deficiency in a brain chemical called acetylcholine, which helps transmit messages between nerve cells. Nefiracetam is a new drug that stimulates acetylcholine. This study will test whether Nefiracetam can safely improve memory, thinking and activities of daily living in patients with mild to moderate intellectual impairment due to Alzheimer's disease.

Patients in the study must have a caregiver and designated representative. Candidates will be given a medical history and physical examination that includes a complete neurologic and neuropsychologic evaluation, blood tests, and an electrocardiogram. A chest X ray and magnetic resonance imaging (MRI) test will be done on patients who have not had these tests within the previous two years. During the 20-week study, each patient will take three pills twice a day for twenty weeks of either Nefiracetame or placebo (sugar pill). Neither the patients nor the doctors will know which patients are getting the drug and which are getting the placebo. Blood and urine tests will be done frequently throughout the study. Patients will be asked to have a spinal tap (on a voluntary basis) to measure the levels of drug in the spinal fluid, and a PET scan (a brain imaging test).

At the end of the study, patients who feel they are doing well with no side effects from the drug (or placebo) may be given the option of continuing treatment for another seven months.

Animal studies showed that Nefiracetam improved learning impairment and memory in rats with dementia. In a small study of humans, about one-fourth of patients who were given a low dose of the drug had improved intellectual function, and about one-half who received a higher dose improved.

DETAILED DESCRIPTION:
Diminished cholinergic function has long been implicated in the pathophysiology of Alzheimer type dementia. Studies in animal models of this disorder as well as in patients with Alzheimer's disease (AD) suggest that drugs capable of activating central cholinergic transmission can improve cognitive function. Nevertheless, no currently available drug of this or any other type consistently confers clinically significant benefit. To further evaluate the cholinergic hypothesis for symptom palliation with a mechanistically novel pharmacologic tool, the acute safety and antidementia efficacy of nefiracetam will be studied using a double-blind, placebo-controlled, parallel groups design. In contrast to the currently available cholinesterase inhibitors, nefiracetam enhances the activity of nicotinic acetylcholine receptors by interacting with a protein kinase C pathway and accelerates acetylcholine turnover and release. Efficacy in patients with mild to moderate dementia will be assessed through application of standardized neuropsychological test instruments in this first double-blind, randomized controlled trial of nefiracetam in AD. Safety will be monitored by means of frequent clinical evaluations and laboratory tests.

ELIGIBILITY:
Study subjects will satisfy NINCDS-ADRDA criteria for probable AD. Dementia severity will be in the mild to moderate range, as evidenced by a Mini-Mental State Examination total score of 12-25 which is roughly equivalent to Alzheimer's Disease Assessment Scale Cognitive (ADAS-Cog) scores of 30 to 11, will include deficits in at least 2 areas of cognition, will have been present at least 1 year, and will have progressed gradually since onset. Patients must be between the ages of 50-90 with onset of dementia after age 40. The modified Hachinski Ischemia Score must be less than 4 and the brain MRI within 2 years of enrollment must be consistent with the diagnosis of AD.

Patients must have had a brain MRI since the onset of dementia symptoms that is consistent with the diagnosis of AD.

Patients must have an acceptable nutritional status (i.e., body weight within 20% of desirable weight for height).

Patients must be surgically sterile.

Patients must be post-menopausal or practicing adequate contraception.

Physical and laboratory exams must be normal, or the abnormalities must be attributed to the dementing illness or judged clinically unimportant to the safe conduct of this trial.

Chest X-ray within 1 year of enrollment must show no active disease.

No history or clinical diagnosis of stroke within 1 year before or concurrent with onset of dementia; hydrocephalus, subdural hematoma, or mass lesion on screening MRI; current seizure disorder; head trauma with loss of consciousness and hospitalization within 1 year before or concurrent with onset of dementia; dementia onset within 1 year following cardiac arrest or surgery; Parkinson's disease (onset prior to or concurrent with dementia), Wilson's, Huntington's, Creutzfeldt-Jakob disease, Pick's disease, or Wernicke's encephalopathy; chronic CNS infection (positive RPR and/or FTA-ABS acceptable if luetic brain disease excluded by documented studies and/or treatment).

No COPD or asthma requiring hospital treatment within 1 year before enrollment (treatment of acute respiratory infections is acceptable).

No acute systemic infection.

No hypothyroidism (TSH greater than 6.0 mclU/ml).

No folic acid (less than 0.9 ng/ml) or B12 deficiency (less than 100 pg/ml) within 1 year before study enrollment.

No recent or acute HAV or HBV infection, or chronic HBV infection by immuno-assays.

No insulin dependent diabetes or poorly controlled non-insulin dependent diabetes.

No history of leukopenia, neutropenia, or thrombocytopenia, cancer (except treated, non-recurrent skin cancer) within 2 years before enrollment.

No severe renal insufficiency (Clcr less than 25 ml/min, BUN greater than 30 mg/dl, or creatinine greater than 2.0 mg/dl), hepatic insufficiency (as indicated by: ASAT (SGOT) 3 x ULN, ALAT (SGPT) 3 x ULN, or total bilirubin greater than 2.0 mg/dl).

No homocysteinemia (greater than 14 micromol/L).

No past history of schizophrenia.

No substance use disorder within 1 year of dementia onset.

No depression requiring medical treatment within the past 30 days.

No administration of tacrine (Cognex) or donezepil (Aricept), investigational drugs, or nutritional supplements used as neurotransmitter precursors for cognitive enhancement within 30 days before enrollment.

No use of anticonvulsants, psychostimulants, centrally acting anticholinergics and agents known to inhibit or be metabolized by CYP 3A4 (e.g., erythromycin, chlarythromycin, troleandomycin, fluconazole, miconazole, ketoconazole, itraconazole and grapefruit juice) within 2 weeks prior to enrollment.

No hepatic, cardiovascular, gastrointestinal, or hematological illness which could interfere with drug absorption, distribution, metabolism, or excretion.

No medical condition that contraindicates cholinergics.

No known hypersensitivity to nefiracetam.

Must be able to swallow/retain tablets.

No history of medical noncompliance.

Must have significant other person or caregiver to assure compliance.

No uncorrectable loss of hearing or eyesight that precludes psychometric testing.

Ability to comprehend instructions or respond to test items of the ADAS and Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) during baseline administration.

No male patients interested in conceiving children given the potential adverse effects on spermatogenesis.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50
Dates: Start 1999-07; Study Completion 2002-01

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States

REFERENCES:
- [Background] Morris JC, Rubin EH. Clinical diagnosis and course of Alzheimer's disease. Psychiatr Clin North Am. 1991 Jun;14(2):223-36. PMID 2062717
- [Background] Henderson AS. Epidemiology of dementia disorders. Adv Neurol. 1990;51:15-25. No abstract available. PMID 2294654
- [Background] Price DL. New perspectives on Alzheimer's disease. Annu Rev Neurosci. 1986;9:489-512. doi: 10.1146/annurev.ne.09.030186.002421. PMID 3518588